CLINICAL TRIAL: NCT03476928
Title: An Open-label, Parallel-group, Randomized, Multicenter Study to Assess the Safety and Efficacy of Vilaprisan in Japanese Subjects With Uterine Fibroids and Heavy Menstrual Bleeding
Brief Title: A Study to Assess the Safety and Efficacy of Vilaprisan in Japanese Subjects With Uterine Fibroids and Heavy Menstrual Bleeding
Acronym: ASTEROID 8
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19435
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Uterine Fibroids and Heavy Menstrual Bleeding
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — vilaprisan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group A1 (Experimental): 4 treatment periods of 12 weeks, each separated by 1 bleeding episode
  Interventions: Drug: Vilaprisan (BAY1002670)
- Treatment Group A2 (Experimental): 2 treatment periods of 24 weeks, separated by 2 bleeding episodes
  Interventions: Drug: Vilaprisan (BAY1002670)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — 2mg, once daily, oral

SUMMARY:
To evaluate the safety and efficacy of vilaprisan in Japanese subjects with uterine fibroids and heavy menstrual bleeding (HMB).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening
* Heavy menstrual bleeding (HMB) >80.00 mL associated with uterine fibroid(s)
* Good general health
* Normal or clinically insignificant cervical smear
* An endometrial biopsy performed during the screening period, without significant histological disorder
* Use of an acceptable nonhormonal method of contraception starting at Visit 1 until the end of the study

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drug
* Any condition requiring immediate blood transfusion
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Abuse of alcohol, drugs, or medicines (e.g., laxatives)
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse event | Up to one year and 3 months

SECONDARY OUTCOMES:
Number of bleeding days | Up to one year and 3 months

CONTACTS AND LOCATIONS:
Locations (25):
- Japan (25):
  - Meitetsu Hospital, Nagoya, Aichi-ken
  - Kano's Clinic for Women, Nagoya, Aichi-ken
  - Kyoritsu Narashinodai Hospital, Funabashi, Chiba
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Jusendo Geneal Hospital Yuasa Foundation, Kōriyama, Fukushima
  - Sato Hospital, Takasaki, Gunma
  - Hashimoto Clinic, Sapporo, Hokkaido
  - Yoshio Clinic, Sapporo, Hokkaido
  - Asahi-Clinic., Takamatsu, Kagawa-ken
  - Kurashiki Medical Clinic, Kurashiki, Okayama-ken
  - Medical Topia Soka Hospital, Sōka, Saitama
  - Sei Womens Clinic, Bunkyo, Tokyo
  - St.Luke's International Hospital, Chuoku, Tokyo
  - Akazawa Clinic, Fuchū, Tokyo
  - Toranomon Womens Clinic, Minato, Tokyo
  - Akasakamitsuke Miyazaki Obstetrics and Gynecology Clinic, Minato, Tokyo
  - Yokokura Clinic, Minato-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Kato Internal medicine and Gynecology Clinic, Fukui
  - Hamanomachi Hospital, Fukuoka
  - Medical corporation keizukai Chayamachi Ladies Clinic, Osaka
  - Medical Corporation Koshinkai Nomura Clinic Namba, Osaka
  - Izuma Clinic, Osaka
  - Shizuoka Saiseikai General Hospital, Shizuoka
  - Toyama Prefectural Central Hospital, Toyama

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, time point and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Momoeda M, Faustmann T, Groettrup-Wolfers E, Kondo M, Yasuda M, Seitz C. Safety and efficacy of vilaprisan in Japanese women with fibroids: The Phase 3 ASTEROID 8 trial. Womens Health (Lond). 2025 Jan-Dec;21:17455057251378954. doi: 10.1177/17455057251378954. Epub 2025 Oct 8. PMID 41059527
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/